CLINICAL TRIAL: NCT01358695
Title: Clinical Trial To Evaluate ANT-1207 In Subjects With Lateral Canthal Lines
Brief Title: Clinical Trial To Evaluate ANT-1207 In Subjects With Crow's Feet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterios Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANT-1207-201-LCL
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Lateral Canthal Lines; Crow's Feet
Keywords: Lateral Canthal Lines; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo Comparator (Placebo Comparator)
  Interventions: Biological: ANT-1207; Biological: Botulinum Toxin Type A
- Dose 1 (Experimental): Dose 1
  Interventions: Biological: ANT-1207; Biological: Botulinum Toxin, Type A; Biological: Botulinum Toxin Type A
- Dose 2 (Experimental): Dose 2
  Interventions: Biological: ANT-1207; Biological: Botulinum Toxin, Type A; Biological: Botulinum Toxin Type A
- Dose 3 (Experimental): Dose 3
  Interventions: Biological: ANT-1207; Biological: Botulinum Toxin, Type A; Biological: Botulinum Toxin Type A
- Dose 4 (Experimental): Dose 4
  Interventions: Biological: Botulinum Toxin, Type A; Biological: Botulinum Toxin Type A
- Dose 5 (Experimental): Dose 5
  Interventions: Biological: Botulinum Toxin, Type A; Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: ANT-1207 — The interventions differ by dose of investigational product applied.
  Arms: Dose 1; Dose 2; Dose 3; Placebo Comparator
Biological: Botulinum Toxin, Type A — The interventions differ by dose of investigational product applied.
  Arms: Dose 1; Dose 2; Dose 3; Dose 4; Dose 5
Biological: Botulinum Toxin Type A — The interventions differ by dose of investigational product applied.

SUMMARY:
The purpose of this study is to provide evidence of the safety, tolerance, and efficacy of ANT-1207 in the treatment of Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate Crow's Feet wrinkles (IGA 2-3) at rest
* moderate to severe Crow's Feet (IGA 3-4) on contraction
* willingness to refrain from any product affecting skin remodeling
* female subjects must be not pregnant and non-lactating

Exclusion Criteria:

* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by Investigator's Global Assessment Score | 2 weeks
  Wrinkle scale with definitions of severity

SECONDARY OUTCOMES:
Subject Self Assessment (SSA) scale | 2 Weeks
  Change from Baseline in the Subject Self Assessment scale
Investigator Global Assessment scale | Week 1, 2, 4, 8, 12
  Change from Baseline in wrinkle scale assessment at all other timepoints

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Baumann Cosmetic & Research Institute, Miami Beach, Florida
  - Palm Beach Esthetic Dermatology and Laser Center, West Palm Beach, Florida
  - William Coleman III, MD, APMC, Metairie, Louisiana
  - Gramercy Park Dermatology, New York, New York
  - Cary Skin Care, Cary, North Carolina